CLINICAL TRIAL: NCT02088957
Title: A Randomized, Open-label, Multicenter, Parallel-group, Exploratory Study to Evaluate the Efficacy of Intravenous Brivaracetam and Intravenous Phenytoin in Subjects Experiencing Nonconvulsive Electrographic Seizures
Brief Title: Efficacy Evaluation of Intravenous Brivaracetam and Phenytoin in Subjects With Nonconvulsive Electrographic Seizures
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termination of study due to low enrollment. There were no safety issues.
Sponsor: UCB BIOSCIENCES, Inc. (Industry)
Collaborators: PRA Health Sciences (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N01394
Expanded Access: NCT03532516 (Available)
Record Dates: First submitted 2014-02-20; First posted 2014-03-17 (Estimated); Results first posted 2016-04-13 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2016-07

CONDITIONS: Nonconvulsive Electrographic Seizures
Keywords: Brivaracetam; Phenytoin; Nonconvulsive electrographic seizures
MeSH Terms: interventions — brivaracetam; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brivaracetam (Experimental): Subjects will receive an acute intravenous (iv) dose of Brivaracetam (BRV) 200 mg as a bolus on Day 1. If seizures recur, a second iv bolus of BRV 100 mg can be given no sooner than 15 minutes after the first bolus. If the second acute bolus is not needed within12 hours after first iv bolus, BRV will be continued as 100 mg iv dose every 12 hours (bid). The total dose for the first 24 hours of treatment should not exceed a maximum dose of 400 mg. The rate of bolus administration is 50 mg (5 mL) undiluted BRV/min. On study Day 5 (or earlier), subjects will transition from iv to oral formulation, at comparable dosing for a maximum of 6 months.
  Subjects should transition to oral medication as soon as they are able to swallow tablets.
  Interventions: Drug: Brivaracetam intravenous solution; Drug: Brivaracetam oral tablets
- Phenytoin (Active Comparator): Subjects will receive an acute intravenous (iv) dose of Phenytoin (PHT) 20 mg/kg at a rate of 50 mg/min on Day 1. If seizures recur, a second acute dose of PHT iv will be given no sooner than 15 minutes after the first dose. Treatment with PHT iv will be continued with at least 2 daily divided doses according to site practice. Daily PHT dose can be adapted according to investigator's clinical judgment. On study Day 5 (or earlier), subjects will transition from iv to oral formulation at comparable dosing for a maximum of 6 months.
  Subjects should transition to oral medication as soon as they are able to swallow tablets.
  Interventions: Drug: Phenytoin intravenous solution; Drug: Phenytoin oral tablets

INTERVENTIONS:
Drug: Brivaracetam intravenous solution — * Active Substance: Brivaracetam
  * Pharmaceutical Form: Solution for infusion
  * Concentration: 10 mg/mL
  * Route of Administration: Intravenous bolus use
  Arms: Brivaracetam
Drug: Brivaracetam oral tablets — * Active Substance: Brivaracetam
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 10 mg and 25 mg tablets; Daily Dose: 200 mg/day (100 mg bid)
  * Route of Administration: Oral use
  Arms: Brivaracetam
Drug: Phenytoin intravenous solution — * Active Substance: Phenytoin
  * Pharmaceutical Form: Solution for infusion
  * Concentration: 50 mg/mL
  * Route of Administration: Intravenous use
  Arms: Phenytoin
Drug: Phenytoin oral tablets — * Active Substance: Phenytoin
  * Pharmaceutical Form: Tablet
  * Concentration: Weight based
  * Route of Administration: Oral use
  Arms: Phenytoin

SUMMARY:
The primary objective of this study is to compare the efficacy of Brivaracetam and Phenytoin, both administered intravenously, in adult subjects experiencing nonconvulsive electrographic seizures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥16 years. Subjects under 18 years may only be included where legally permitted and ethically accepted
* Subjects in the neurological intensive care unit (NICU) (or equivalent closely monitored environment) having brain insult including traumatic brain injury and having nonconvulsive electrographic seizures (NCES) confirmed by electroencephalogram (EEG), lasting a minimum of 10 seconds but not >30 minutes (minimum of 1 seizure in the last 6 hours) and treatment with an antiepileptic drug (AED) is required according to the physician's clinical judgment
* Subject is expected to be under cEEG monitoring with video surveillance in the Neuro ICU for at least 36 hours from the first administration of study drug

Exclusion Criteria:

* Subject has history of severe adverse hematologic or cutaneous reaction to any drug
* Subject presenting with status epilepticus or nonconvulsive status epilepticus (NCSE) (ie, 1 continuous, convulsive or nonconvulsive, unremitting seizure lasting >30 minutes during Visit 1)
* Subject has been diagnosed with anoxic brain injury
* Subject has a known history of status epilepticus during the 6 months preceding Visit 1
* Subject is currently treated with Levetiracetam (LEV) or Phenytoin (PHT) or has been treated within the last 30 days before Visit 1 with LEV or PHT
* Subject is on felbamate with <18 months' exposure before Visit 1
* Subject has presence of any sign (clinical or imaging techniques) suggesting a rapidly progressing process such that the subject is not expected to survive >48 hours
* Subject has any clinical condition that would impair reliable participation in the study or necessitate the use of medications not allowed by the protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (2):
- United States (2):
  - 3, Lexington, Kentucky
  - 1, Jackson, Mississippi

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty subjects were planned to be screened in order to enroll 50 subjects in a 1:1 ratio to intravenous (iv) Brivaracetam (BRV) or iv Phenytoin (PHT) with stratification based on categorized age (<65 years versus ≥65 years) across approximately 15 sites.
Pre-assignment Details: This study was stopped due to low enrollment; the termination date was 17 Nov 2014. One subject enrolled, but discontinued from the study prematurely due to lack of efficacy.
Period: Overall Study
Arm/Group | Brivaracetam | Phenytoin
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Population: Demographics of the only subject included are presented below.
Arm/Group | Brivaracetam
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Seizure Freedom for 12 Hours Based on cEEG/vEEG Monitoring Which Starts 1 Hour After the End of the Last Acute iv Administration of Study Drug and Prior to the Initiation of Bid (Twice a Day) Dosing
Description: Seizure freedom is based on cEEG/vEEG (continuous video electroencephalogram) monitoring.
Time Frame: From 1 hour after end of the last acute iv administration of study drug and prior to initiation of bid dosing (which begins 12 hours after the last acute iv administration of study drug)
Population: This variable was not analyzed and no results are available.
Arm/Group | Brivaracetam | Phenytoin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Percentage of Subjects With Seizure Freedom for 12 Hours Based on cEEG/vEEG Monitoring Which Starts After the End of the Last Acute Intravenous (iv) Administration of Study Drug and Prior to the Initiation of Bid (Twice a Day) Dosing
Description: Seizure freedom is based on cEEG/vEEG (continuous video electroencephalogram) monitoring.
Time Frame: From end of the last acute iv administration of study drug and prior to initiation of bid dosing (which begins 12 hours after the last acute iv administration of study drug)
Population: This variable was not analyzed and no results are available.
Arm/Group | Brivaracetam | Phenytoin
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Time to Achievement of 12 Hours of Seizure Freedom Relative to the Start of the First Acute Intravenous (iv) Administration
Description: Seizure freedom is based on cEEG/vEEG (continuous video electroencephalogram) monitoring.
Time Frame: From start of first acute iv administration on Day 1
Population: This variable was not analyzed and no results are available.
Arm/Group | Brivaracetam | Phenytoin
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Achievement of 12 Hours of Seizure Freedom Relative to the Start of the Last Acute Intravenous (iv) Administration That Occurred Prior to the Initiation of Bid (Twice a Day) Dosing
Description: Seizure freedom is based on cEEG/vEEG (continuous video electroencephalogram) monitoring.
Time Frame: From start of last acute iv administration prior to initiation of bid dosing (which begins 12 hours after the last acute iv administration of study drug)
Population: This variable was not analyzed and no results are available.
Arm/Group | Brivaracetam | Phenytoin
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Percentage of Subjects Requiring a Second Acute Intravenous (iv) Administration Between 15 Minutes to 12 Hours After First Acute iv Administration
Time Frame: Between 15 minutes to 12 hours after first acute iv administration
Population: This variable was not analyzed and no results are available.
Arm/Group | Brivaracetam | Phenytoin
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Time to First Onset of Seizure Cessation Relative to the Start of the First Acute Intravenous (iv) Administration
Description: Seizure cessation is based on cEEG/vEEG (continuous video electroencephalogram) monitoring.
Time Frame: From start of first acute iv administration
Population: This variable was not analyzed and no results are available.
Arm/Group | Brivaracetam | Phenytoin
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events were collected during the 75 days the only subject was included in this study.
Description: Adverse Events of the only subject included are presented below.
Arm/Group | Brivaracetam | Phenytoin
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (N=1) | Phenytoin (N=0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Decreased urinary output (Investigations) | 1 (1) | 0 (0)
iv infiltration (General disorders) | 1 (1) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days